CLINICAL TRIAL: NCT04541030
Title: UAB-NCI Collaborative Study on Integrating Genomic Prostate Score With MRI Targeted Prostate Biopsies
Brief Title: Integrated Genomic Prostate Score With MRI Targeted Prostate Biopsies
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920136; 20-C-N136
Record Dates: First submitted 2020-09-05; First posted 2020-09-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Prostate Cancer
Keywords: Gleason Score; Multiparameter MRI; Focal Therapy; Natural History
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GPS Cohort 1: Samples and images from up to 277 evaluable patients diagnosed with NCCN low or intermediate risk prostate cancer, Gleason <= 7, managed with RP, and mpMRI within 6 months prior to prostatectomy

SUMMARY:
Background:

Prostate cancer is one of the most common cancers in men. For some men, their cancer is monitored. Others have surgery to remove the prostate. Focal therapy is another treatment option. It treats the areas of cancer selectively, which leaves the rest of the prostate intact. This can help lessen side effects. Men who get focal therapy must be chosen carefully. The Oncotype DX Genomic Prostate Score (GPS) assay tests biopsy samples for certain cancer-related genes. It then then gives a score from 1 to 100 to predict the likelihood of poor outcomes. The GPS is used to choose men for focal therapy. Researchers want to test the GPS further.

Objective:

To assess how GPS may be useful when used with MRI to improve how men are chosen for focal therapy of prostate cancer.

Eligibility:

Men age 18 and older who had NCCN low or intermediate risk prostate cancer and had MRI and radical prostatectomy at the Urologic Oncology Branch, National Cancer Institute and collaborating centers.

Design:

This is a multisite study. It will review data and samples that were collected in the past. Samples and images from up to 277 participants will be used.

Tumor tissue will be tested with the GPS.

Data such as age at diagnosis, race, biopsy results, and pathology results will be merged with the GPS results.

Data will be entered into an in-house electronic system. It will be password protected. All data will be kept in secure sites that comply with NIH security standards.

DETAILED DESCRIPTION:
Background:

* Prostate cancer is one of the most common malignancies occurring in men. While many men will qualify for active surveillance (AS), those with intermediate risk disease are often recommended definitive therapy despite the morbidity.
* Focal therapy for prostate cancer has been promoted as an alternative to the standard paradigm of immediate radical prostatectomy (RP) versus AS for prostate cancer management. Focal therapy treats the areas of cancer selectively, leaving the remainder of the prostate intact.
* While focal therapy offers great promise in terms of minimizing side effects and helping prostate cancer patients avoid radical therapies, careful patient selection is required.
* The Oncotype DX Genomic Prostate Score (GPS) assay was developed using the ability to extract and amplify RNA of sufficient quantity and quality from the very small amounts of prostate tumor tissue from biopsy samples. Using these samples, a discovery study identified 12 cancerrelated genes associated with multiple clinically relevant endpoints including adverse pathology, biochemical recurrence, clinical recurrence, and prostate cancer associated death.
* The GPS assay uses these 12 genes and 5 reference genes to construct an algorithm giving a score from 0-100 to predict the likelihood of adverse pathology.
* The goal of this study is to evaluate how GPS may be useful in conjunction with MRI to improve patient selection for focal therapy of prostate cancer.

Objectives:

-To determine if there is a positive association between continuous GPS score and occult high risk and/or non-organ confined disease on whole mount prostatectomy specimens where an MRI was performed less than 6 months before diagnostic biopsy, and the biopsy was less than 6 months before RP and the lesion was not identified on multiparameter MRI (mpMRI)

Eligibility:

* Samples and images from men, over 18 years old, who were diagnosed with NCCN low or intermediate risk prostate cancer and were managed with radical prostatectomy at the Urologic Oncology Branch, National Cancer Institute and collaborating centers
* Biopsy Gleason Score <= 7
* Multiparametric MRI, with images available for review, within 6 months prior to the prostatectomy
* Availability of adequate diagnostic biopsy tissue specimen for GPS analysis

Design:

* This multisite study will be a prospective analysis of retrospective data.
* Samples and images will be obtained from will consist of approximately 277 evaluable patients who were diagnosed with NCCN low or intermediate risk prostate cancer and were managed with RP at the Urologic Oncology Branch, National Cancer Institute and collaborating centers.
* In the interest of a demographically diverse cohort, samples and images from patients from UAB will be identified, working in reverse chronological order until the cohort is complete or eligible specimens are exhausted; remaining cases will then be selected from the NCI patient population, also working in reverse chronological order.
* Tumor tissue from the highest-grade lesion will be tested with the Oncotype DX Genomic Prostate Scor for generation of the GPS.
* Clinical characteristics including but not limited to age at diagnosis, race, PSA, biopsy results, Prostate MRI PIRADS score, and surgical pathology results will be collected and merged with GPS results.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Samples and images from men > =18 with NCCN very low, low, or intermediate risk prostate cancer with tumor tissue that meet the pathologic tissue requirements of the Oncotype DX Genomic Prostate Score assay
* Biopsy Gleason Score 7 or lower within 6 months preceding radical prostatectomy
* 3Tesla MRI with/without coil performed within 6 months preceding diagnostic biopsy
* Availability of diagnostic biopsy

EXCLUSION CRITERIA:

* Any active therapy received for prostate cancer (e.g., hormonal treatment, radiation, chemotherapy, biologic agents, surgery) prior to radical prostatectomy. 5 alpha reductase inhibitor treatment will not be considered to be hormonal treatment for this definition
* Men with NCCN high risk or very high-risk prostate cancer
* Biopsy Gleason 8
* No biopsy tissue available
* Missing surgical pathology whole mount, or unwilling to send surgical pathology whole mount to NCI for review
* Missing diagnostic PSA
* Missing clinical T stage
* Known lymph node positive or metastatic disease at time of diagnosis
* Missing MRI 6 months before diagnostic biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from male patients with NCCN low or intermediate risk disease managed with radical prostatectomy (multiparametric MRI (mpMRI) performed within 6 months prior to the prostatectomy indicating localized, organ confined disease and adequate diagnostic biopsy tissue specimen).
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
relationship between continuous GPS score and occult high-risk disease | 2-3 years
  To determine if there is a positive relationship between continuous GPS score and occult high-risk disease on whole mount prostatectomy specimens where an MRI was performed less than 6 months before diagnostic biopsy, and the biopsy was less than 6 months before RP and the lesion was not identified on mpMRI

SECONDARY OUTCOMES:
distributions of clinical, pathological and demographic variables | 2-3 years
  To compare the distributions of clinical, pathological and demographic variables for the Genomic Health, Inc. (GHI) study cohort with all the eligible samples from patients in the participating institutions databases

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - National Cancer Institute (NCI), Bethesda, Maryland